CLINICAL TRIAL: NCT00674050
Title: A Phase 1, Open-Label Study to Investigate the Effect of Albuterol (Salbutamol) and Fluticasone on the Pharmacokinetics of Inhaled Technosphere® Insulin Inhalation Powder in Healthy Subjects
Brief Title: A Study Designed to Determine if the Drugs Albuterol (Salbutamol) and Fluticasone Have an Effect on the Pharmacokinetics of the Investigational Product Technosphere® Insulin Inhalation Powder in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-114
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes Mellitus; Healthy Subjects
Keywords: Healthy Males or Females subjects
MeSH Terms: conditions — Diabetes Mellitus | interventions — Albuterol; Fluticasone

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Technosphere Insulin (TI) Inhalation Powder; Drug: Albuterol (Salbutamol); Drug: Fluticasone

INTERVENTIONS:
Drug: Technosphere Insulin (TI) Inhalation Powder — 3.0 U of human insulin. 5 or 10 mg or Technosphere Inhalation Powder, containing 15 0r 30 U of insulin.
Drug: Albuterol (Salbutamol) — 2 puff= 200ug total dose
Drug: Fluticasone — 2 puffs= 500ug total dose

SUMMARY:
This study will investigate the effects of inhaled albuterol & fluticasone on one dose of TI Inhalation Powder. A total of 12 eligible subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Subjects must have a fasting blood glucose (BG) level of less than 6.1 mmol/L FEV1/ FVC = LLN TLC = 80% Predicted DLco (unc) = 80% Predicted (Miller) No significant improvement in pre- to post-bronchodilator spirometry (defined as an increase of = 12% and = 200 mL in FEV1 or FVC) at Screening FEV1 = 80% (NHANES III Predicted

Exclusion Criteria:

History of diabetes mellitus Previous exposure to any inhaled insulin product Any known pulmonary disease or inability to perform PFT maneuvers meeting recommended American Thoracic Society (ATS) standards of acceptability and repeatability criteria Respiratory tract infection within 8 weeks prior to Screening/Visit 1 Major organ system diseases including seizures, heart failure, uncontrolled hypertension, aneurysm, cancer within the past 5 years, liver disease, anemia or autoimmune disorder Clinically significant abnormalities on screening laboratory evaluation Female subjects who are pregnant, lactating, or planning to become pregnant during the clinical trial period or not practicing adequate birth control Unable and/or unlikely to comprehend how to use the investigational device in this study or to follow study instructions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
PK parameters of serum insulin | 0-360 min

CONTACTS AND LOCATIONS:
Overall Officials: Anders H. Boss, Study Chair — Mannkind Corporation
Locations (1):
- ICON Development Solutions, Manchester, United Kingdom, United Kingdom